CLINICAL TRIAL: NCT07163806
Title: Diagnostic Value of Volumetric Parameters of 18F-FDG PET/CT in Characterizing Thyroid Incidentalomas.
Brief Title: Volumetric Parameter of 18F-FDG PET/CT in Characterizing Thyroid Incidentalomas
Status: Not yet recruiting | Type: Observational
Sponsor: Fatma Abelzaher Mahmoud Ahmed (Other)
Responsible Party: Sponsor-Investigator, Fatma Abelzaher Mahmoud Ahmed, fatma abdelzaher, Assiut University
Organization: Assiut University (Other)
Other Study IDs: thyroid incidentaloma PET/CT
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Incidentalomas
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET/CT with 18-FDG — Patients will fast for at least four hours before imaging with blood glucose level <200 mg /dL before intravenous administration of about 3.7 MBq/kg (0.1 mCi/kg). Imaging will be performed approximately 45 to 60 min after 18F-FDG injection , an imaging field of view from the base of skull to mid thighs with the arms above the head whenever possible is used or otherwise the arms are positioned beside the body.
  The semiquantitative analysis will be done using standardized uptake values (SUV). The SUV calculation will be done via the default method by body weight [(SUV = mean ROI activity (MBq/g)/injected activity (MBq)/body weight (g)]. For measurement of SUVs of lesion, multiple circular ROIs will be drawn covering the lesion over its entire length. For healthy organs, a circular ROI of 10 mm diameter will be drawn

SUMMARY:
To assess the clinical significance of FDG-avid thyroid incidentalomas detected on PET/CT and explore correlations between SUV max, ultrasound characteristics, and histopathology for suspicious lesion.

DETAILED DESCRIPTION:
Thyroid incidentalomas are unsuspected thyroid lesions discovered during imaging performed for unrelated medical reasons. With the expanding use of 18F-fluorodeoxyglucose positron emission tomography/computed tomography (18F-FDG PET/CT) for cancer staging and follow-up, the detection of incidental thyroid nodules particularly those showing focal FDG uptake-has significantly increased (Are C et al., 2007; Kim TY et al.,2005). Although the overall prevalence of thyroid incidentalomas detected on PET/CT is relatively low (reported between 1.1% and 4%), the risk of malignancy among FDG-avid nodules is high, ranging from 26.7% to 64.6%, which is considerably greater than in non-FDG-avid nodules (Shi H et al.,2018; Makis W & Ciarallo A, 2017;Choi JY et al., 2006).

Globally, thyroid cancer is one of the most common endocrine malignancies, with an increasing incidence rate over the past two decades (Sung H et al.,2021). In Egypt, recent data indicate that thyroid cancer accounts for approximately 2.6% of all new cancers, with a noticeable increase in detection largely attributed to the rise in imaging investigations (Ibrahim AS et al., 2014;GLOBOCAN, 2020). Despite this increase, clinical guidelines still lack aconsensus on how to best manage thyroid incidentalomas detected by PET/CT, especially in resource-limited settings.

Previous studies have explored various semi-quantitative PET parameters, particularly SUVmax, as potential indicators of malignancy. Malignant thyroid incidentalomas tend to show significantly higher SUVmax values than benign ones, but considerable overlap exists, limiting its standalone diagnostic value (Shi H et al., 2018; Kim BH et al., 2013).

Furthermore, integrating ultrasound characteristics such as microcalcifications, hypoechogenicity, irregular margins, and taller-than-wide shape, has shown promise in enhancing diagnostic accuracy (Haugen BR etal., 2016; Russ G et al., 2017). However, data on how well these PET/CT and ultrasound features correlate with final histopathology remain limited in Egypt and other low-resource settings.

In a large meta-analysis, the pooled risk of malignancy in FDG-avid thyroid incidentalomas was estimated at 34.6% (Bertagna F et al., 2012), but single-center studies report wide variability, which may be due to differences in patient selection, imaging thresholds, and follow-up protocols. Given the growing detection of FDG-avid thyroid nodules and the lack of clear, standardized management protocols in Egypt, there is a critical need for localized research to guide decision-making and reduce unnecessary surgeries or missed malignancies

ELIGIBILITY:
Inclusion Criteria:

* All Adult patients referred for 18F-FDG PET/CT and found to have thyroid incidentalomas,

Exclusion Criteria:

* o Known history of thyroid malignancy.

  * Previous thyroid surgery .

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All Adult patients referred for 18F-FDG PET/CT and found to have thyroid incidentalomas,
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Assess the clinical significance of FDG-avid thyroid incidentalomas on PET/CT | 3 years
  Assess the clinical significance of FDG-avid thyroid incidentalomas on PET/CT and explore correlations between SUVmax, TIRAD system on ultrasound, and final histopathology for suspicious lesion.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Achury C, Estorch M, Domenech A, Camacho V, Flotats A, Jaller R, Geraldo L, Deportos J, Montes A, Carrio I. [Interpretation of thyroid incidentalomas in (18)F-FDG PET/CT studies]. Rev Esp Med Nucl Imagen Mol. 2014 Jul-Aug;33(4):205-9. doi: 10.1016/j.remn.2013.12.006. Epub 2014 Feb 21. Spanish. PMID 24560597